CLINICAL TRIAL: NCT03588962
Title: RESTenosis in Patients With Contact ALLergy to Metals Zabrze Study
Brief Title: Metal Allergy In-Stent Restenosis Study
Acronym: RESTALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Mariusz Gasior, Professor of Medicine, Head of III Dept. of Cardiology, Silesian Centre for Heart Diseases
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RESTALL Zabrze Study
Record Dates: First submitted 2018-03-18; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Metal Allergy; Contact Allergy; Restenoses, Coronary; In-stent Restenosis; Coronary Artery Disease
Keywords: allergy to metals, restenosis, in-stent restenosis; coronary artery disease
MeSH Terms: conditions — Dermatitis, Allergic Contact; Coronary Restenosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metal allergy driven restenosis (Experimental): Patients with angiographically proven in-stent restenosis developed after technically correct implantation. Patch tests for the metals used in stent production will be applicated. The tests will be applicated during the hospitalisation, then read after 48 hours and 72 hours, and subsequently interpreted by the skilled dermatologist, during the hospital stay or afterwards. Possible correlation between allergy to metals utilised during the stent manufacturing (nickel, cobalt, chromium, molybdenum, tungsten) and in-stent restenosis occurence.
  Interventions: Biological: In-stent restenosis
- Looking for allergic restenosis (Placebo Comparator): Patients with (technically correctly) implanted stent. Patch tests will be applicated to identify cases with contact allergy. The tests will be applicated during the hospitalisation, then read after 48 hours and 72 hours, and subsequently interpreted by the skilled dermatologist, during the hospital stay or afterwards.The patients will then be monitored for a 12 months follow-up period in purpose of evaluating the dependance between in-stent restenosis and contact allergy. Possible correlation between allergy to metals utilised during the stent manufacturing (nickel, cobalt, chromium, molybdenum, tungsten) and in-stent restenosis occurence.
  Interventions: Biological: In-stent restenosis

INTERVENTIONS:
Biological: In-stent restenosis — Patch tests for the metals applicated in each of the patients

SUMMARY:
In-stent restenosis remains one of the most challenging problems in patients after coronary artery angioplasty. Angiographically, it is discovered in 10% of the patients after drug-eluting stent (DES) implantation. There are multiple factors causing restenosis, which can be divided into two major groups: first vessel-dependent (based on the vessel's tortuosity, dimensions and lesion's calcification, all leading to suboptimal stent expansion), and second dependent on the inflammatory processes caused by the intervention. Study objectives is the analysis of the possible correlation between allergy to metals utilised during the stent manufacturing (nickel, cobalt, chromium, molybdenum, tungsten) and in-stent restenosis occurence. The angiographic results of stent implantation, and in-stent restenosis will be assessed independently by two skilled interventional cardiologists, and in case of their discrepant opinions, the decision will be made on the basis of the third cardiologist. The tests will be applicated during the hospitalisation, then read after 48 hours and 72 hours, and subsequently interpreted by the skilled dermatologist, during the hospital stay or afterwards.

DETAILED DESCRIPTION:
Introduction:

In-stent restenosis remains one of the most challenging problems in patients after coronary artery angioplasty. Angiographically, it is discovered in 10% of the patients after drug-eluting stent (DES) implantation. There are multiple factors causing restenosis, which can be divided into two major groups: first vessel-dependent (based on the vessel's tortuosity, dimensions and lesion's calcification, all leading to suboptimal stent expansion), and second dependent on the inflammatory processes caused by the intervention. Although the proper stent expansion depends mostly on the cardiologist's manual dexterity, the inflammation development does totally not depend on the operator. The allergic reactions to metals are likely to be one of the underlying causes of inflammation. Among the most prevalent allergens, cobalt, chromium, nickel, and tungsten used as the stent materials are causing the most intensive contact allergic reaction. The allergic process induced by the aforementioned metals belongs to type IV contact allergy (T-cell mediated). Stent implantation results in life-long contact with metal, thus in allergic patients, it is likely to develop local reactions leading to in-stent restenosis. Up to date, there have been approximately one thousand in-stent restenosis cases documented in patients with confirmed contact allergy to stent metals.

Study objectives:

Analysis of the possible correlation between allergy to metals utilised during the stent manufacturing (nickel, cobalt, chromium, molybdenum, tungsten) and in-stent restenosis occurence.

Materials and methods:

The study will consist of two arms:

First arm: Patch tests for the metals used in stent production will be applicated in the patients with angiographically proven in-stent restenosis developed after technically correct implantation.

Second arm: In patients with (technically correctly) implanted stent, patch tests will be applicated to identify cases with contact allergy. The patients will then be monitored for a 6-12 months follow-up period in purpose of evaluating the dependance between in-stent restenosis and contact allergy.

The angiographic results of stent implantation, and in-stent restenosis will be assessed independently by two skilled interventional cardiologists, and in case of their discrepant opinions, the decision will be made on the basis of the third cardiologist.

The tests will be applicated during the hospitalisation, then read after 48 hours and 72 hours, and subsequently interpreted by the skilled dermatologist, during the hospital stay or afterwards.

ELIGIBILITY:
Inclusion Criteria:

* angiographically proven in-stent restenosis after technically correct implantation
* technically correctly implanted stent

Exclusion Criteria:

* autoimmune diseases (e.g., rheumatoid arthritis)
* immunodeficiency syndromes (e.g., HIV infection)
* chronic use of immunosuppressive drugs and/or corticosteroids
* skin lesions that may attenuate the reading of skin tests
* previous coronary artery bypass surgery (in subgroup 1) or planned coronary artery bypass surgery (in subgroup 2)
* any surgical procedure with metal implants (in the past or planned within 12 months of observation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 12 months
  In-stent restenosis, acute myocardial infarction (AMI), death, cardiovascular (CV) death

IPD SHARING:
Plan to Share IPD: No